CLINICAL TRIAL: NCT00480883
Title: Treatment of Cutaneous Leishmaniasis With Meglumine Antimoniate 20 Mg/Kg/Day Versus Meglumine Antimoniate 10 Mg/Kg/Day And Tablet Allopurinol 20 Mg/Kg/Day
Brief Title: Treatment of Cutaneous Leishmaniasis With Meglumine Antimoniate Versus Meglumine Antimoniate and Allopurinol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Combined Military Hospital, Pakistan (Other)
Responsible Party: DR AMER EJAZ, COMBINED MILITARY HOSPITAL, KHARIAN, PAKISTAN
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2007-05-29; First posted 2007-05-31 (Estimated); Last update posted 2010-06-02 (Estimated); Status verified 2008-05

CONDITIONS: Leishmaniasis, Cutaneous
Keywords: cutaneous leishmaniasis of the old world
MeSH Terms: conditions — Leishmaniasis, Cutaneous | interventions — Meglumine Antimoniate; Allopurinol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): injection meglumine antimoniate 20 mg/kg/day/intramuscular for 21 days.
  Interventions: Drug: meglumine antimoniate
- 2 (Experimental): injection meglumine antimoniate 10 mg/kg/day/intramuscular plus tablet allopurinol 1200 mg/day/6hourly divided doses.
  Interventions: Drug: meglumine antimoniate, allopurinol

INTERVENTIONS:
Drug: meglumine antimoniate, allopurinol — first drug in injectable, second is in tablet form.
  Arms: 2
Drug: meglumine antimoniate — injectable 20 mg/kg/day/intramuscular for 21 days.
  Arms: 1
Drug: meglumine antimoniate, allopurinol — injectable meglumine antimoniate 10 mg/kg/day/intramuscular for 21 days plus tablet allopurinol 300mg/4times a day for 21 days.
  Arms: 2

SUMMARY:
Background: Cutaneous Leishmaniasis is a worldwide disease, endemic in over 88 countries, that has shown an increasing incidence over the last many decades. For the last 60 years antimony compounds are considered the treatment of choice. Though their use is expensive, cumbersome, has many adverse effects and not effective in all patients, the search for a better alternative is still going on. Low dose antimony compounds in combination with several agents have shown promise of reducing adverse effects of antimony compounds without compromising efficacy. Allopurinol is one such agent which though promising lacks randomized, controlled trials to prove efficacy. The main objective of this study is to evaluate low dose sodium stibogluconate in combination with allopurinol and to compare it with high dose sodium stibogluconate in terms of efficacy and adverse effects.

Methods and design: A multi-center randomized, controlled trial including 620 patients from endemic areas for Leishmaniasis in Pakistan will be undertaken to assess the research question. Parasitologically confirmed cutaneous leishmaniasis will be included in the study. After evaluating the inclusion/exclusion criteria patients will be randomized to receive either meglumine antimoniate (20 mg/kg/day/intramuscular, till clinical resolution or a maximum of 28 days) or combination of meglumine antimoniate (10 mg/kg/day intramuscular) and allopurinol (20 mg/kg/day/oral) till clinical resolution or a maximum of 28 days. During treatment patients will be admitted to hospital and monitored daily for the presence of adverse effects. Follow up period will last six months during which patients will visits the research centers for assessment of healing process at monthly intervals.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between 18 and 50 years old.
* Cutaneous ulcers, nodules, plaques, of more than two weeks of evolution requiring systemic therapy.
* Positive parasitological diagnosis for cutaneous leishmaniasis.
* Patients that voluntarily accept to participate in the study and sign the informed consent.
* Disposition to be admitted to hospital, if necessary, and to attend all the visits punctually (initial, treatment and follow up).
* Acceptation of not using any other treatment for cutaneous leishmaniasis while in the study.

Exclusion Criteria:

* Pregnant women.
* Presence of any condition or disease that compromises the patient immunologically (i.e. diabetes, cancer, etc.) or, any other, that, based on the judgment of the researcher, could alter the course of cutaneous leishmaniasis.
* Diffuse cutaneous leishmaniasis.
* Visceral leishmaniasis.
* Complete or incomplete treatment with antimony compounds in the last three months.
* Patients with history of hepatic, renal, or cardiovascular disease.
* Mentally or neurologically disabled patients that are considered not fit to approve their participation in the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2008-01; Primary Completion 2008-06 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
clinical healing of lesions. | 3 months

SECONDARY OUTCOMES:
improvement of more than 50% in lesion size | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: AMER EJAZ, FCPS, Principal Investigator — Combined Military Hospital, Pakistan
Locations (1):
- Combined Military Hospital, Kharian Cantonment, Punjab Province, Pakistan

REFERENCES:
- [Background] Momeni AZ, Reiszadae MR, Aminjavaheri M. Treatment of cutaneous leishmaniasis with a combination of allopurinol and low-dose meglumine antimoniate. Int J Dermatol. 2002 Jul;41(7):441-3. doi: 10.1046/j.1365-4362.2002.01527.x. PMID 12121563